CLINICAL TRIAL: NCT04113928
Title: Maximising the Bioavailability and Activity of Broccoli Phytochemicals Using a Broccoli Soup Enriched for Myrosinase by Addition of Mustard Seeds
Brief Title: Broccoli Ileo Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: University of Reading (Other); The James Hutton Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 14/SC/1326
Record Dates: First submitted 2019-09-17; First posted 2019-10-03 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Ileostomy - Stoma
Keywords: Broccoli; Bioavailability; Ileostomists; Randomised controlled trial; Phytochemical

STUDY DESIGN:
Intervention Model Description: Randomised double blind crossover design.
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Broccoli & mustard seed soup (Experimental): 200ml acute feed
  Interventions: Dietary Supplement: Broccoli & mustard seed soup; Dietary Supplement: Broccoli soup
- Broccoli soup (Active Comparator): 200ml acute feed
  Interventions: Dietary Supplement: Broccoli & mustard seed soup; Dietary Supplement: Broccoli soup

INTERVENTIONS:
Dietary Supplement: Broccoli & mustard seed soup — 200ml acute feed
Dietary Supplement: Broccoli soup — 200ml acute feed

SUMMARY:
Epidemiological and experimental studies have indicated that the consumption of diets rich in cruciferous vegetables such as broccoli has a range of beneficial effects on human health. These effects are usually attributed to naturally-occurring glucosinolates and their breakdown products, isothiocyanates, in cruciferous vegetables. One of these compounds, sulforaphane, the hydrolysis product of glucoraphanin, the main glucosinolate in broccoli has been reported to have bactericidal activity against H. pylori and other human pathogens. The investigators have recently shown that adding mustard seeds, which contain a more resilient form of this enzyme, to processed broccoli actually increased the formation of sulforaphane and minimised production of another biologically-inactive form. Experimental studies by the investigators have shown that sulforaphane can inhibit growth of a number of enteric pathogens including salmonella and E. coli which exert their effects in the small intestine. Currently the bioavailability, stability and bioactivity of sulforaphane in the small intestine of a human following consumption of broccoli is not known.

To assess the effect of broccoli phytochemicals in vivo 20 participants who have previously had an ileostomy (removal of colon, > 1.5 years post operative) will be fed 200 ml of broccoli soup/control in a randomised double blind crossover design and collect the ileal fluid before (0 hr) and after (4 hr) the feeding. The ileal fluid collected from participants will have undergone in vivo digestion, allowing analysis of the chemical composition and bioactivity of the ileal fluid. The hypothesis to be tested is that consumption of cooked broccoli plus myrosinase from mustard seeds will result in high levels of sulforaphane in ileostomy fluid, sufficient to suppress growth of enteric pathogens. This study will be used to assess whether previous observations on the in vitro antibacterial activity of broccoli are relevant in vivo.

ELIGIBILITY:
Inclusion Criteria:

* undergone an ileostomy and be more than 1.5 year post-operative
* non smoking

Exclusion Criteria:

* not undergone an ileostomy and/or is less than 1.5 year post-operative
* smoker.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-03-23 (Actual); Primary Completion 2015-04-03 (Actual); Study Completion 2015-04-03 (Actual)

PRIMARY OUTCOMES:
Phytochemical concentration | Change over 4 hours
  Ileal fluid analysis by Gas Chromatography Mass Spec (GCMS) and Liquid Chromatography / Mass Spec (LC/MS)

SECONDARY OUTCOMES:
Inhibition of enteric pathogens | Change over 4 hours
  Ileal fluid tissue culture analysis (zone of inhibition (mm))

CONTACTS AND LOCATIONS:
Locations (1):
- Human Intervention Studies Unit, Ulster University, Coleraine, Co.Londonderry, United Kingdom

IPD SHARING:
Plan to Share IPD: No